CLINICAL TRIAL: NCT03343977
Title: A Prospective Open-label, Randomized, Two-arm Pilot Study to Investigate the Toxicity and Pharmacokinetics of 2-Weekly and 3-Weekly Docetaxel in Metastatic Hormone-Sensitive Prostate Cancer.
Brief Title: Toxicity & Pharmacokinetics of 2 & 3-weekly Docetaxel in Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn for technical reasons
Sponsor: Peng Wang, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Peng Wang, MD PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17-GU-71
Record Dates: First submitted 2017-10-06; First posted 2017-11-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Every two weeks docetaxel (Experimental): 50 mg/m2 of docetaxel will be given on day 1 every 14 days over one hour IV infusion for up to 9 cycles (1 cycle = 14 days)
  Interventions: Drug: docetaxel 50mg/m2
- Every three weeks docetaxel (Active Comparator): 75 mg/m2 of docetaxel will be given on day 1 every 21 days over one hour IV infusion for up to 6 cycles (1 cycle = 21 days)
  Interventions: Drug: docetaxel 75mg/m2

INTERVENTIONS:
Drug: docetaxel 50mg/m2 — 50 mg/m2 of docetaxel will be given on day 1 every 14 days
  Arms: Every two weeks docetaxel
Drug: docetaxel 75mg/m2 — 75 mg/m2 of docetaxel will be given on day 1 every 21 days
  Arms: Every three weeks docetaxel

SUMMARY:
This study is designed to investigate the toxicity and pharmacokinetics (PK) of 2-weekly and 3-weekly docetaxel in metastatic hormone-sensitive prostate cancer (mHSPC). Also, a mechanism-based population pharmacokinetics/pharmacodynamics (PK/PD) model will be developed to provide a better understanding of the complex relationships between the drug exposure and toxicity profiles of docetaxel in mHSPC.

DETAILED DESCRIPTION:
This pilot study is designed to investigate the toxicity and PK of 2-weekly and 3-weekly docetaxel in mHSPC. Furthermore, a mechanism-based population PK/ pharmacodynamics (PD) model will be developed to provide a better understanding of the complex relationships between the drug exposure and toxicity profiles of docetaxel in mHSPC. In addition, selected pro-inflammatory and macrophage-associated cytokines will be collected to assess the potential role of these cytokines as the early markers of docetaxel resistance in patients with mHSPC. (Cytokines: macrophage inhibitory cytokine 1 (MIC1), interleukin (IL)-1ra, IL-1β, IL-4, IL-6, IL-12, and IFNγ). Serological response, defined as a prostate-specific antigen (PSA) level of <0.2 ng/mL at 12 months, and progression-free survival at 12 months are selected as the secondary clinical endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed prostate cancer with EXTENSIVE metastatic disease and have been on androgen deprivation therapy for <90 days. Hormonal therapy must not have commenced more than 90 days prior to study.

   Definition of extensive disease: Metastases involving at least one lesion in any bony structures beyond the vertebral column and pelvic bone or any involvement with viscera. In the absence of visceral lesion, there must be four or more bone lesions. Patients with disease limited to vertebral column and/or pelvis alone with or without lymph node or lymph node only disease involvement are not eligible for this trial.
2. Age ≥18 years.
3. ECOG performance status ≤2 (Karnofsky ≥60%).
4. Patients must have normal organ and marrow function as defined below within four weeks prior to the study:

   * Absolute neutrophil count ≥1,500/mcL
   * Platelets ≥100,000/mcL
   * Total bilirubin less than ULN
   * AST(SGOT)/ALT(SGPT) ≤1.5 × institutional upper limit of normal
   * Alkaline phosphate ≤2.5 x ULN
   * Creatinine clearance ≥ 30 mL/min calculated using the Cockcroft-Gault formula: Creatinine clearance for male (mL/min) = (140-age)*(body weight in kg)/(72 x serum creatinine in mg/dl)
5. If a patient has had major surgery, the patient must be longer than four weeks post surgery and must have recovered from all toxicity prior to beginning protocol study.
6. Peripheral neuropathy with Grade ≤1
7. Patients may be enrolled if they have had prior palliative radiation therapy. However, this has to have been commenced within 30 days of starting androgen deprivation.
8. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who are receiving any other investigational agents.
2. Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
3. History of hypersensitivity to docetaxel or polysorbate 80.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social dysfunction that could impair the ability of the patients to participate in the study or interfere with interpretation of study results.
5. Docetaxel is a CYP3A4 substrate and caution should be taken with its use and any drugs known to interact with it. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference for this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Appendix B contains a list of known drugs that are contraindicated or have major interactions with docetaxel.
6. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with docetaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
7. Patients with prior docetaxel chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-14 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the neutropenia toxicity rate over time between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | Baseline; at each therapy cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen); at 6-, 9-, and 12-months post treatment
  Toxicity rate in each arm will be estimated based on a one-sided 90% confidence interval. Assuming at most a 31% neutropenia rate, a sample of 16 patients per arm will provide a one-sided 90% confidence interval upper limit equal to 50%.

SECONDARY OUTCOMES:
Comparison of the pharmacokinetics (PK) parameter 'Cmax' (maximum concentration) between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | 0, 0.25, 0.75, 3, 6.5, and 24 hours post first docetaxel infusion; and, at the end of docetaxel infusion of the last cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen)
  Individual docetaxel PK parameters will be estimated by non-compartmental method using Phoenix WinNonlin software (Certara Corporation, Princeton, NJ). Maximum concentration (Cmax) will be the observed value.
Comparison of the pharmacokinetics (PK) parameter 'Tmax' (time to Cmax) between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | 0, 0.25, 0.75, 3, 6.5, and 24 hours post first docetaxel infusion; and, at the end of docetaxel infusion of the last cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen)
  Individual docetaxel PK parameters will be estimated by non-compartmental method using Phoenix WinNonlin software (Certara Corporation, Princeton, NJ). Time to Cmax (Tmax) will be the observed value.
Comparison of the pharmacokinetics (PK) parameter 'AUClast' between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | 0, 0.25, 0.75, 3, 6.5, and 24 hours post first docetaxel infusion; and, at the end of docetaxel infusion of the last cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen)
  Area under the plasma concentration-time curve from zero to last observed time (AUClast) will be estimated using the trapezoidal rule.
Comparison of the pharmacokinetics (PK) parameter 't1/2' (terminal half-life) between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | 0, 0.25, 0.75, 3, 6.5, and 24 hours post first docetaxel infusion; and, at the end of docetaxel infusion of the last cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen)
  Terminal half-life (t1/2) will be calculated using the terminal linear portion of the log concentration-time curve.
Comparison of the pharmacokinetics (PK) parameter 'AUC0-inf' (area under the curve from zero to infinity)' between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | 0, 0.25, 0.75, 3, 6.5, and 24 hours post first docetaxel infusion; and, at the end of docetaxel infusion of the last cycle (a cycle is 2 weeks for the 2-weekly regimen, 3 weeks for the 3-weekly regimen)
  AUC from zero to infinity (AUC0-inf) will be determined using the following equation:
  AUC0-inf = AUClast + Cllast/Kel Where Clast is the observed concentration at the last time point and Kel is the slope of the terminal linear portion of the log concentration-time curve.
Comparison of all grades of neutropenia (including febrile neutropenia) and other toxicities between the 2-weekly docetaxel dosing regimen and the 3-weekly docetaxel dosing regimen in metastatic hormone-sensitive prostate cancer. | up to 12 months after the first docetaxel dose
  Adverse event data and corresponding toxicity grades during the days of treatment will be summarized for each docetaxel dosing arm. Neutropenia rates will be estimated along with exact 90% one-sided binomial confidence intervals. Incidence, frequency, severity, and attribution tables for other toxicities will be generated.
Development of a population system pharmacology model to describe the relationships between the PK (drug exposure) and PD (toxicity) of 2-weekly docetaxel in metastatic hormone-sensitive prostate cancer | CBC with differential and platelet will be collected: 24-hour +/- 3hrs; and 7 days +/- 1day after the first administration of 2-weekly docetaxel in cycle 1 to support the development of population PK/PD model
  The mechanism population PK/PD model will be developed using Monte-Carlo Expectation-Maximization algorithm implemented S-ADAPT software (version 1.57, BMSR, Log Angeles, CA).
Development of a population system pharmacology model to describe the relationships between the PK (drug exposure) and PD (toxicity) of 3-weekly docetaxel in metastatic hormone-sensitive prostate cancer | CBC with differential and platelet will be collected: 24-hour +/- 3hrs; 7 days +/- 1day; and 14 days +/- 1day after the first administration of 3-weekly docetaxel in cycle 1 to support the development of population PK/PD model
  The mechanism population PK/PD model will be developed using Monte-Carlo Expectation-Maximization algorithm implemented S-ADAPT software (version 1.57, BMSR, Log Angeles, CA).
Evaluation of the rate of complete serological response at 12 months | 12 months post treatment
  Defined as a prostate-specific antigen (PSA) level of less than 0.2 ng/mL
Evaluation of the cytokine profile before and after treatment at different docetaxel dosage regimens | Baseline before chemotherapy; immediately prior to second dose (cycle length depends on dosing regimen) of chemotherapy; 30 minutes prior to chemotherapy at Week 7, and at Week 19; at Month 12 after start of first docetaxel dose.
  Descriptive statistics will be calculated for each cytokine parameter measured at each time point for each docetaxel dosing regimen and comparison from pre vs post-treatment within each arm will be performed using paired t-test while comparisons of cytokine parameters between docetaxel dosing groups will likewise be performed using two-sample t-test. Several cytokine parameters are evaluated and we will employ the Holm's p-value adjustment method to account for multiple testing between dosing group arms.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States